CLINICAL TRIAL: NCT03654924
Title: Continuous Laryngeal Cuff Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSRB 2016/00604
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2018-08

CONDITIONS: Value of Continuous Pressure Monitoring in Laryngeal Mask
Keywords: LMA; Leak; Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Observational study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laryngeal Mask (Experimental): A pressure gauge will be connected to the LMA using a small cable to measure the LMA cuff pressure continuously.
  Interventions: Device: Laryngeal Mask

INTERVENTIONS:
Device: Laryngeal Mask — General anaesthesia using LMA will be performed as per standard procedure. A pressure gauge will be connected to the LMA using a small cable to measure the LMA cuff pressure continuously.

SUMMARY:
The aim of this study is to evaluate the airway seal of LMA during intraoperative manipulation.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) is widely used in dental surgery as it provides an unobstructed airway and provides a reliable seal from bleeding and surgical debris. However, there have been few studies of the integrity of the LMA seal during intraoperative surgical manipulation with the use of the LMA.

In general anesthesia using LMA, airway and esophagus cannot be separated completely. Insufficient airway seal become the risk of aspiration in airway management. This study will focus on airway seal following LMA use in dental surgery.

ELIGIBILITY:
Inclusion Criteria:

* NUH patients who will undergo wisdom teeth extraction.

Exclusion Criteria:

* Patients with tooth braces
* Patients who are at risk of aspiration
* Patients with missing any of incisor tooth
* Pregnant woman
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Utility of continuous LMA cuff pressure monitoring in dental surgery | Intra-operatively
  Measure of intra cuff pressure

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, MBBS, MMed, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, results, analysis